CLINICAL TRIAL: NCT03175640
Title: Implementation to Motivate Physician Response to Opioid Dependence in HIV Settings
Brief Title: Prescribe to Save Lives
Acronym: PTSL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baystate Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); The Miriam Hospital (Other); Boston Medical Center (Other); Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Peter Friedmann, Chief Research Officer and Endowed Chair for Clinical Research, Baystate Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: BH-15-259; R01DA038082 (NIH)
Record Dates: First submitted 2017-05-18; First posted 2017-06-05 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Opioid-Related Disorders; Drug Overdose
MeSH Terms: conditions — Opioid-Related Disorders; Drug Overdose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implementation intervention (Experimental)
  Interventions: Behavioral: Implementation intervention

INTERVENTIONS:
Behavioral: Implementation intervention — The implementation intervention includes peer-to-peer training, post-training outreach, proactive expert support, and assistance with addressing environmental barriers.

SUMMARY:
The U.S. is in the midst of an epidemic of opioid overdose deaths. The common use of opioids among persons living with HIV, along with their common use of benzodiazepines, has resulted in high rates of opioid overdose among this population. This study will test the implementation of evidence-based training, mentoring, technical support, and academic detailing to encourage HIV physicians to adopt evidence-based interventions to reduce overdose risk and treat opioid addiction.

ELIGIBILITY:
Inclusion Criteria:

Clinicians and staff of HIV practice sites that:

* Receive Ryan White Funding;
* Treat adults with HIV;
* Have 3 or more prescribing clinicians;
* Have an electronic medical record (EMR) with an electronic medication list.

Exclusion Criteria:

* Sites located in states with fewer than 500 Persons Living With HIV (PLWH) will be excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in naloxone prescribing behavior | baseline to 6 months
  Number of clinicians that prescribe naloxone. This information will be collected from electronic medical record (EMR) data.

SECONDARY OUTCOMES:
Change in perception about pharmacotherapy for opioid use disorder; 6-month | baseline to 6 months
  Opinions About Medication Assisted Treatment (OAMAT) survey
Change in perception about pharmacotherapy for opioid use disorder; 12-month | baseline to 12 months
  Opinions About Medication Assisted Treatment (OAMAT) survey
Change in prescribing motivation; 6 months | baseline to 6 months
  Change in Motivation Scale
Change in prescribing motivation; 12 months | baseline to 12 months
  Change in Motivation Scale
Change in prescriber training | baseline to 12 months
  Number of prescribers that have completed buprenorphine training.
Change in buprenorphine prescribing behavior | baseline to 12 months
  Prevalence of buprenorphine prescription. This information will be collected from EMR data.

CONTACTS AND LOCATIONS:
Overall Officials: Peter D Friedmann, MD, MPH, Principal Investigator — University of Massachusetts Medical School - Baystate; Josiah D Rich, MD, MPH, Principal Investigator — The Miriam Hospital
Locations (2):
- United States (2):
  - University of Massachusetts Medical School - Baystate, Springfield, Massachusetts
  - The Miriam Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
The investigators will make study data available to the community of scientists and the public in keeping with NIDA policies. After all data have been collected and the results of the major papers are in press, de-identified data will be made available to other qualified researchers on request. The request will be evaluated by Dr. Friedmann to ensure that it meets reasonable standards of scientific integrity. Ultimately, it is anticipated that de-identified data and codebooks will be warehoused and available through the ICPSR and SAMHDA websites. This data sharing plan will comply with the requirements of the privacy rule and federal regulations under HIPAA and 42 CFR Part 2 that govern the protection of individually identifiable information.

REFERENCES:
- [Derived] Jawa R, Walley AY, Wilson DJ, Green TC, McKenzie M, Hoskinson R Jr, Bratberg J, Ramsey S, Rich JD, Friedmann PD. Prescribe to Save Lives: Improving Buprenorphine Prescribing Among HIV Clinicians. J Acquir Immune Defic Syndr. 2022 Aug 15;90(5):546-552. doi: 10.1097/QAI.0000000000003001. PMID 35587832